CLINICAL TRIAL: NCT02507661
Title: Esthetic Outcomes of Implant-supported Crowns After Alveolar Ridge Preservation With Beta Tricalcium Phosphate and Collagen in the Maxillary Esthetic Zone
Brief Title: Effect of Alveolar Ridge Preservation on Implant Esthetic Outcomes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Belgrade (Other)
Responsible Party: Principal Investigator, Bozidar Brkovic, DDS, MSc, PhD, Professor, DDS PhD Professor, University of Belgrade
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 36/21
Record Dates: First submitted 2015-06-11; First posted 2015-07-24 (Estimated); Last update posted 2018-03-23 (Actual); Status verified 2018-03

CONDITIONS: Partial Edentulism
MeSH Terms: interventions — beta-tricalcium phosphate; Collagen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- alveolar ridge preservation - 2 months (Experimental): preservation of alveolar ridge with beta tricalcium phosphate + collagen - 2 months
  Interventions: Drug: preservation of alveolar ridge with beta tricalcium phosphate + collagen - 2 months
- no-preservation of alveolar ridge - 2 months (Active Comparator): no-preservation of alveolar ridge - 2 months
  Interventions: Drug: no-preservation of alveolar ridge - 2 months
- preservation of alveolar ridge - 4 months (Experimental): preservation of alveolar ridge with beta tricalcium phosphate + collagen - 4 months
  Interventions: Drug: preservation of alveolar ridge with beta tricalcium phosphate + collagen - 4 months
- no-preservation of alveolar ridge - 4 months (Active Comparator): no-preservation of alveolar ridge - 4 months
  Interventions: Drug: no-preservation of alveolar ridge - 4 months
- preservation of alveolar ridge - 9 months (Experimental): preservation of alveolar ridge with beta tricalcium phosphate + collagen - 9 months
  Interventions: Procedure: preservation of alveolar ridge with beta tricalcium phosphate + collagen - 9 months
- no-preservation of alveolar ridge - 9 months (Active Comparator): no-preservation of alveolar ridge - 9 months
  Interventions: Drug: no-preservation of alveolar ridge - 9 months

INTERVENTIONS:
Drug: preservation of alveolar ridge with beta tricalcium phosphate + collagen - 2 months
  Arms: alveolar ridge preservation - 2 months
Drug: no-preservation of alveolar ridge - 2 months
  Arms: no-preservation of alveolar ridge - 2 months
Drug: preservation of alveolar ridge with beta tricalcium phosphate + collagen - 4 months
  Arms: preservation of alveolar ridge - 4 months
Drug: no-preservation of alveolar ridge - 4 months
  Arms: no-preservation of alveolar ridge - 4 months
Procedure: preservation of alveolar ridge with beta tricalcium phosphate + collagen - 9 months
  Arms: preservation of alveolar ridge - 9 months
Drug: no-preservation of alveolar ridge - 9 months
  Arms: no-preservation of alveolar ridge - 9 months

SUMMARY:
The purpose of this study is to evaluate esthetic outcome of implant supported single crowns after alveolar ridge preservation with beta three calcium phosphate with collagen type I in aesthetic region in upper jaw.

ELIGIBILITY:
Inclusion Criteria:

* healthy patients according to Classification of American Society of Anesthesiologists (ASA I)
* presence of 4 socket walls
* non-smokers
* good oral hygiene
* good occlusion

Exclusion Criteria:

* patients with alveolar ridge height less than 12 mm
* presence of acute or chronic oro-facial pain
* acute periapical infection
* injured soft tissue
* patients who had dental interventions in last 7 days
* patients who had any medications within last 24 hours
* patients with bruxism and para-functions
* patients with allergies to any of applied materials

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
implant stability analysis at the time of implant placement | baseline
  Implant stability will be measured by the resonance frequency analysis
implant stability analysis 3 weeks after implant placement | baseline, 3 weeks
  Implant stability will be measured by the resonance frequency analysis
implant stability analysis 6 weeks after implant placement | baseline, 6 weeks
  Implant stability will be measured by the resonance frequency analysis
implant stability analysis 8 weeks after implant placement | baseline, 8 weeks
  Implant stability will be measured by the resonance frequency analysis
change in pink and white esthetic score 2 months of loading | 2 months
  Pink esthetic scale and white esthetic scale will be used for evaluation of changes in white and pink esthetic parameters for implant-supported crowns
change in pink and white esthetic score 6 months of loading | 6 months
  Pink esthetic scale and white esthetic scale will be used for evaluation of changes in white and pink esthetic parameters for implant-supported crowns
change in pink and white esthetic score 12 months of loading | 12 months
  Pink esthetic scale and white esthetic scale will be used for evaluation of changes in white and pink esthetic parameters for implant-supported crowns

SECONDARY OUTCOMES:
analysis of new bone formation 2 months after preservation of alveolar ridge | 2 months
  New bone formation will be assessed by histological analysis and histomorphometrical measurement
analysis of new bone formation 4 months after preservation of alveolar ridge | 4 months
  New bone formation will be assessed by histological analysis and histomorphometrical measurement
analysis of new bone formation 9 months after preservation of alveolar ridge | 9 months
  New bone formation will be assessed by histological analysis and histomorphometrical measurement

CONTACTS AND LOCATIONS:
Overall Officials: Bozidar M Brkovic, PhD, Principal Investigator — School of Dental Medicine, University of Belgrade
Locations (1):
- School of Dental Medicine, University of Belgrade, Belgrade, Serbia